CLINICAL TRIAL: NCT03956966
Title: Ultrasound-guided Quadratus Luborum Block Using Bupivacaine Versus Bupivacaine-Dexamethasone for Postoperative Analgesia in Laparoscopic Cholecystectomy
Brief Title: Quadratus Luborum Block Using Bupivacaine Versus Bupivacaine-Dexamethasone in Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, haidy salah mansour, principle investigator, Minia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 88-11/2018
Record Dates: First submitted 2019-05-08; First posted 2019-05-21 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Post Operative Pain
Keywords: Quadratus Lumborum Block; Laparoscopic Cholecystectomy; dexamethasone
MeSH Terms: conditions — Pain, Postoperative | interventions — Sodium Chloride; Bupivacaine; Dexamethasone

STUDY DESIGN:
Intervention Model Description: randomized, double blind
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- saline (Placebo Comparator): bilateral quadratus lumborum block using 0.9% normal saline
  Interventions: Drug: TQL block with saline
- Bupivacaine (Active Comparator): bilateral quadratus lumborum block using Bupivacaine hydrochloride 0.25%
  Interventions: Drug: TQL block with Bupivacaine
- Bupivacaine and dexamethasone (Active Comparator): bilateral quadratus lumborum block using Bupivacaine hydrochloride 0.25% and dexamethasone
  Interventions: Drug: TQL block with Bupivacaine and dexamethasone

INTERVENTIONS:
Drug: TQL block with saline — drug: saline 21 ml 0.9% normal saline administered on each side as bilateral TQL blocks Drug: fentanyl With induction of general anaesthesia, fentanyl (1 microgram.kg) will be given. Intraoperatively, fentanyl boluses (0.5 microgram.kg) will be given in case of increase in intraoperative mean arterial blood pressure or heart rate of more than 20% of baseline for longer than 5 minutes.
  Drug: Paracetamol Paracetamol infusion (15 mg.kg) will be given by intravenous infusion after induction of general anesthesia. Postoperatively, 1 g of paracetamol will be given by intravenous infusion to all cases every 8 hours.
  Drug: Ketorolac analgesia In PACU Ketorolac 30 mg ampoule will be given by intravenous infusion to all cases Drug: Nalbuphine Nalbuphine boluses 0.1 mg. /kg will be given as rescue analgesia if VAS is more than3.
  Device: ultrasound-guided nerve block Transmuscular quadratus lumborum block, ultrasound-guided
  Other Names: C Group
  Arms: saline
Drug: TQL block with Bupivacaine — Drug: saline
  1mL 0.9% normal saline administered on each side as bilateral TQL blocks drug: Bupivacaine 20 ml Bupivacaine hydrochloride 0.25% administered on each side as bilateral TQL blocks Drug: fentanyl With induction of general anaesthesia, fentanyl (1 microgram.kg) will be given. Intraoperatively, fentanyl boluses (0.5 microgram.kg) will be given in case of increase in intraoperative mean arterial blood pressure or heart rate of more than 20% of baseline for longer than 5 minutes.
  Drug: Paracetamol 15 mg.kg will be given by intravenous infusion after induction of general anesthesia. Postoperatively, 1 g of paracetamol will be given to all cases every 8 hours.
  Drug: Ketorolac In PACU Ketorolac 30 mg ampoule will be given by intravenous infusion to all cases Drug: Nalbuphine Nalbuphine boluses 0.1 mg. /kg will be given as rescue analgesia if VAS is more than 3.
  Device: ultrasound-guided nerve block Transmuscular quadratus lumborum block
  Other Names: B Group
  Arms: Bupivacaine
Drug: TQL block with Bupivacaine and dexamethasone — Drug: dexamethasone
  1 mL dexamethasone "4mg" administered on each side as bilateral TQL blocks drug: Bupivacaine 20 ml Bupivacaine hydrochloride 0.25% administered on each side as bilateral TQL blocks Drug: fentanyl With induction of general anaesthesia, fentanyl (1 microgram.kg) will be given. Intraoperatively, fentanyl boluses (0.5 microgram.kg) will be given in case of increase in MBP or HR of more than 20% of baseline for longer than 5 minutes.
  Drug: Paracetamol Paracetamol infusion (15 mg.kg) will be given by intravenous infusion after induction of general anesthesia. Postoperatively, 1 g of paracetamol will be given by intravenous infusion to all cases every 8 hours.
  Drug: Ketorolac In PACU Ketorolac 30 mg ampoule will be given by intravenous infusion to all cases Drug: Nalbuphine Nalbuphine boluses 0.1 mg. /kg will be given as rescue analgesia if VAS is more than 3.
  Device: ultrasound-guided nerve block Transmuscular quadratus lumborum block
  Other Names: D Group
  Arms: Bupivacaine and dexamethasone

SUMMARY:
The aim of the present study was to compare the effectiveness of transmuscular Quadratus Lumborum block using Bupivacaine versus Bupivacaine- Dexamethasone in providing analgesia in patients undergoing laparoscopic cholecystectomy.

Because postoperative pain after laparoscopic surgery is complex, specialists suggest that effective analgesic treatment should be a multimodal support. Quadratus lumborum block (QLB) is a new abdominal truncal block for controlling somatic pain in both the upper and lower abdomen. Dexamethasone, through its anti-inflammatory and blocking effects on neural discharge, and nociceptor C fibers transmission could be used as a local anesthetic adjuvant.

DETAILED DESCRIPTION:
The patients were randomly allocated into three groups each contains (30) patient. Control group (C) received bilateral ultrasound guided quadratus lumborum block using (20 ml 0.9% normal saline + 1mL 0.9% normal saline) in each side ,Bupivacaine group (B) received bilateral quadratus lumborum block using (20 ml Bupivacaine hydrochloride 0.25% + 1mL 0.9% normal saline) in each side and Dexamethasone-Bupivacaine group (D) received bilateral quadratus lumborum block using (20 ml Bupivacaine hydrochloride 0.25% + 1 mL dexamethasone "4mg") in each side.

The following variables: heart Rate, mean arterial Blood Pressure, peripheral oxygen saturation, visual analogue pain scale , time to first analgesic request, total Analgesic requirement in the first 24 hours, patient satisfaction and complications were Recorded and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* American Physical Status I or II
* Elective laparoscopic Cholecystectomy

Exclusion Criteria:

* Patient refusal.
* Hematological diseases
* Bleeding disorders.
* Coagulation abnormality.
* Psychiatric diseases.
* Local skin infection
* Sepsis at site of the block.
* Known intolerance to the study drugs.
* Body Mass Index > 40 Kg/m2.
* Emergency laparoscopic cholecystectomy
* If laparoscopic procedure converted to open.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Time for first request to rescue analgesia | 24 hours
  Time for the first request to rescue analgesia (in minutes)

SECONDARY OUTCOMES:
postoperative Nalbuphine | 24 hours after surgery
  Cumulative postoperative Nalbuphine consumption (total dose given in milligrams)
intraoperative fentanyl | For 4 hours after start of anaesthesia
  Cumulative intraoperative fentanyl consumption (total dose given in micrograms)
Postoperative pain severity will be assessed using VAPS | For 24 hours after surgery
  The severity of postoperative pain will be measured and recorded by using the visual analogue scale (VAPS) for pain, where 0 is equal to no pain and 10 indicates the worst possible pain
side effects | For 24 hours after surgery
  Incidence of postoperative nausea and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Haidy S Mansour, MD, Study Director — assistant professor of Anesthesia and Surgical Intensive Care
Locations (1):
- Minya University, Minya, Egypt